CLINICAL TRIAL: NCT01386099
Title: A Phase IIa Study to Build an Understanding of the Pharmacokinetic-Pharmacodynamic Relationship of PSN821 in Type 2 Diabetes Patients (T2DM).
Brief Title: A PK-PD Study of PSN821 in Type 2 Diabetes Patients (T2DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prosidion Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSN821-202; MCC Trial Reference no (Other: 20110147)
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- PSN821 (Experimental)
  Interventions: Drug: PSN821
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PSN821 — Three PSN821 dose groups: PSN821 75mg twice a day, 250mg twice a day and 625mg twice a day for 12 weeks.
  Arms: PSN821
Drug: Placebo — Placebo twice a day for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics and pharmacodynamics of PSN821 in patients with type 2 diabetes.

Subjects will be assessed for beta-cell function using a hyperglycaemic clamp before the start of treatment and at the end of a 12 week treatment period as the primary endpoint. HbA1c, fasting plasma glucose and body weight are secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes according to the American Diabetes Association criteria, diagnosed at least 12 months prior to screening.
* Male or female, between 18 and 75 years of age, inclusive.
* Body Mass Index of 25 - 45 kg/m2, inclusive.
* Diabetes managed on a stable regimen of diet, exercise and metformin monotherapy (without dosage adjustments within 4 weeks prior to screening).
* Haemoglobin A1c (HbA1c) of 7.5 10% at screening.
* Fasting plasma glucose (FPG) of between 7 - 13.3 mmol/L at screening and Day -1.
* Males who are, and whose partners are able to comply with contraceptive advice.
* Females of non child-bearing potential.
* Willing to sign the written Informed Consent Form (ICF) to participate in the study and to abide by the study restrictions.

Exclusion Criteria:

* Patients with Type 1 diabetes or maturity onset diabetes of the young or secondary forms of diabetes, such as due to pancreatitis.
* Marked diabetic complications.
* Illness or medication that impacts on the scientific integrity of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Beta-cell function | 12 weeks
  Subjects will be assessed for beta-cell function using a hyperglycaemic clamp before the start of treatment and at the end of a 12 week treatment period as the primary endpoint.

SECONDARY OUTCOMES:
HbA1c | 12 weeks
  HbA1c
Fasting plasma glucose | 12 weeks
  Fasting plasma glucose
Body weight | 12 weeks
  Body weight

CONTACTS AND LOCATIONS:
Locations (4):
- South Africa (4):
  - Synexus Clinical Research SA (Pty) Ltd, Pretoria, Gauteng
  - Parexel Bloemfontein, Bloemfontein
  - Parexel George, George
  - Parexel Port Elizabeth, Port Elizabeth